CLINICAL TRIAL: NCT04459689
Title: Worldwide COVID-19 in Children and Adult Patients With Primary ImmunoDeficiencies (PID) Survey
Brief Title: COVID-19 in PID Survey
Acronym: COPID19
Status: Recruiting | Type: Observational
Sponsor: Imagine Institute (Other)
Responsible Party: Sponsor
Other Study IDs: COPID19
Record Dates: First submitted 2020-07-02; First posted 2020-07-07 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Primary Immune Deficiency; COVID
MeSH Terms: conditions — Primary Immunodeficiency Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
With the emergence of SARS-CoV-2 and the COVID-19 pandemic, there is an urgent need to understand the impact of infection on immunodeficient individuals. Whilst co-morbidities (such as diabetes, cancer, arterial hypertension, heart disease...) have been documented in people infected with SARS-CoV-2, there is currently no information on the consequences and outcomes for individuals with primary immunodeficiencies (PID).

Following the 1st phase of the survey (launched by Isabelle Meyts (ESID), Nizar Mahlaoui (CEREDIH & IPOPI) and Kate Sullivan with Stuart Tangye (IUIS), that gave an idea of the number of affected PID patients and the impact of SARS-CoV-2 and directly focusing on obtaining this top level of information), we are launching the 2nd phase: "COPID19".

COPID19 survey is a secured online GDPR compliant platform based in Paris (Imagine Institute). It has been approved by the Paris-Necker-Enfants malades IRB and Ethics Committee. However, this retrospective survey is designed for global distribution. Data can be entered by a health care professional (mostly clinicians) through a personal login and password.

Each documenting person will have access to his/her own patients' data. COPID19 require a greater level of information than the 1st phase. The eCRF will be open to evolutions depending on progresses in our knowledge of this pandemic.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with a Primary Immune Deficiency
* COVID-19 (proven or probable)

Exclusion Criteria:

* Secondary Immune Deficiency
* Other Coronovirus infection

Min Age: 0 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All patients with Primary Immune Deficiency and COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-03-15 (Actual); Primary Completion 2027-02-18 (Estimated); Study Completion 2027-02-18 (Estimated)

PRIMARY OUTCOMES:
Survival of patients with PID affected by COVID-19 | Baseline
Rate of admission to ICU of patients with PID affected by COVID-19 | Baseline
Rate of oxygen therapy of patients with PID affected by COVID-19 | Baseline

SECONDARY OUTCOMES:
Sequelae of patients with PID affected by COVID-19 | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Nizar MAHLAOUI, MD, MPH, PhD, Study Chair — Necker Enfants Malades University Hospital
Locations (1):
- Imagine Institute, Paris, France

IPD SHARING:
Plan to Share IPD: No